CLINICAL TRIAL: NCT02468245
Title: Does a Nursing Intervention Improve Adherence to Oral Chemotherapies in the Outpatient Cancer Treatment Setting?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Kelly Morris, RN, Nurse Manager, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1096
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Antineoplastic Agents
Keywords: Nursing intervention; compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): This is a "usual care" group. Patients in this arm will receive the standard pre-drug initiation training and 4 week clinic follow up visit.
  Interventions: Behavioral: usual care
- Intervention arm (Experimental): Patients in this arm will also receive the standard pre-drug initiation training followed by telephone follow up by an oncology certified chemotherapy nurse (OCN) at week one, two, and three. Patients will then have the standard 4 week follow up clinic visit.
  Interventions: Behavioral: weekly telephone follow up

INTERVENTIONS:
Behavioral: weekly telephone follow up — For the study group, at the initial education visit, a time for each phone call that is convenient for the patient will be scheduled. At each phone call, the OCN will get a pill count and discuss reasons for missed doses if applicable; grade any AE's experienced and interventions for those side effects; and answer any questions or concerns that they patient may be having. Patients will then return for the standard 4 week clinic visit.
  Arms: Intervention arm
Behavioral: usual care — The control group will receive the standard chemotherapy education and will return for the standard 4 week follow up clinic visit.
  Arms: Control Arm

SUMMARY:
This study is being conducted by Bassett Healthcare Network in coordination with Bassett Cancer Institute. Patients prescribed oral chemotherapies will be approached to consider consent to this study. This study will try to establish if nursing interventions can help improve patients' adherence to taking their oral chemotherapies as prescribed by their doctor. Oral chemotherapies are emerging as a growing treatment of choice for many cancer diagnoses. Adherence to the prescribed treatment plan is very important to gain the best response to these types of treatments. The study will examine if nursing intervention via weekly phone calls may help improve adherence to oral chemotherapy treatment plans.

DETAILED DESCRIPTION:
The purpose of this study is to investigate which nursing intervention will help to improve adherence in adult patients who are receiving oral chemotherapy. This study will identify the barriers to adherence, interventions that will increase patients' adherence, and the role of nursing in promoting oral chemotherapy adherence. Oral chemotherapy adherence is important in the setting of cancer care as many new chemotherapy medications being approved for use are oral chemotherapies. Nursing responsibility in this study is to help promote interventions that would improve adherence. The literature shows that the best intervention to promote adherence to oral chemotherapy is education that patients receive prior to them starting their treatment. The interventions such as the MEMS system, AVR, and the generic diary were studied and found to be somewhat effective in improving adherence, but not reliable. The literature supports the use of individualized and personalized education for patients. The education should be in terms that they can understand and absorb, and it should be information that they need related to their treatment.

Oral chemotherapy has emerged as the growing treatment of choice in the cancer treatment specialty; accounting for a quarter of the 400 anticancer medications currently under development (Simchowitz et al., 2010). There are now more than 20 oral antineoplastic agents approved for use in the United States alone; and dozens more under development (Ruddy, Mayer, & Partridge, 2009). Chemotherapy treatments are moving in the direction of conveniences for patients. Oral chemotherapies can be given to patients to take home and be administered in the convenience of their homes. This process works for some patients, but not all.

One of the biggest issues that health care providers find with oral chemotherapy is the non-adherence with the regimens. Without nursing education and follow up interventions, adherence is even more difficult to obtain. Although some patients want to experience having the same care and intervention as a patient receiving intravenous chemotherapy, the mindset of receiving oral chemotherapy is that it is just a pill and not taken seriously by some patients. In a study conducted at Dana Farber, most patients would prefer oral chemotherapy to intravenous (IV) chemotherapy for its convenience, ease of use, and painless administration (Simchowitz et al., 2010). Although most patients realize the importance of taking their medication and adhering to the regimen, they are still non-adherent and suffer unneeded side effects due to that non-adherence. Not to mention that they do not get the full therapeutic effect of the oral chemotherapy regimen.

The standard process for treatment with oral chemotherapy agents start with the providers request for the agent via prescription. Once patient has received approval and has the drug available, the patient will call the cancer center to set up a formal educational appointment with an oncology certified chemotherapy nurse (OCN). The OCN meets with the patient to review potential side effects, how to manage those side effects, and how to properly take the oral chemotherapy. It will be at this education appointment that, the patient will be approached for interest in the study.

Subjects will be identified as any patient that has an oral chemotherapy prescribed that meets the inclusion criteria (please see inclusion/exclusion criteria list later in this document). If the patient expresses interest informed consent process will begin.Once patient has given informed consent, the OCN will confirm eligibility. Once consented and eligibility verified, they will be randomized to either the control group (no intervention, standard of care [SOC]) or to the study group (the intervention group). The initial sample size is 60. All eligible patients' prescribed oral chemotherapy will be approached until sample size of 60 participants has been reached. An interim analysis will be completed after 60 patients have completed the study to assess adequacy of the sample size.

If randomized to the study arm, the OCN will follow-up with that patient at week one, two, three via phone,. At week four, follow-up will occur at the patients routinely scheduled medical oncology visit. For the control group, data will be collected at initial education visit and again at the 4 week physician visit. At the initial education visit both the study group and the control group will receive the standard chemotherapy education, and complete a QOL questionnaire. For the study group, at the initial education visit, a time for each phone call that is convenient for the patient will be scheduled. At each phone call, the OCN will get a pill count and discuss reasons for missed doses if applicable; grade any adverse events (AE's) experienced and interventions for those side effects; and answer any questions or concerns that they patient may be having.

The control group will not receive contact by the OCN at week 1, 2 and 3. At week four, both the control group and the study group will have a complete physical, pill count, QOL completion and document any AE experienced.

The quality of life (QOL) survey tool will be a questionnaire that is self-reported by the patient. This will be done at the initial education session and again at the four week follow up session, for both the control and the intervention group. The sample size will be 60 participants, 30 for the control group and 30 for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Must be >= 18 years of age
* Have a diagnosis of Cancer that will require an oral chemotherapy
* Be treated at Bassett Medical Center Cancer Center
* Must not be receiving radiation or infusional chemotherapy concomitantly with their oral chemotherapy

Exclusion Criteria:

* Being treated at satellite sites
* Receiving radiation and/or infusional chemotherapy concurrently with oral chemotherapy
* Due to impairment or other reasons, patient unable to provide consent or comply with survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Oral chemotherapy compliance | 4 weeks
  A 4 week pill count will be completed on all participants to measure drug compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Loeffler, RN, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States